CLINICAL TRIAL: NCT03122275
Title: Stepwise Strategy to Improve Cervical Cancer Screening Adherence (SCAN-CC): Automatic Text Messages, Phone Calls and Face-to-face Interviews
Brief Title: Stepwise Strategy to Improve CANcer Screening Adherence: Cervical Cancer
Acronym: SCAN-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: João Firmino Domingues Barbosa Machado (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Sponsor-Investigator, João Firmino Domingues Barbosa Machado, Principal Investigator, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EPIUnit_SCANCC_2017
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Mass Screening; Early Detection of Cancer; Uterine Cervical Neoplasm; Text Message; Reminder Systems
Keywords: Adherence; Directive Counseling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepwise intervention (Experimental): Stepwise approach, with increasing complexity and cost, to improve adherence to organized cervical cancer screening, implemented through three steps:
  step 1a - customized text message invitation; step 1b - customized automatic phone call invitation; step 2 - secretary phone call; step 3 - health professional phone call and face-to-face appointment.
  Intervention stops whenever the participant adheres to organized screening or after undergoing the complete stepwise intervention.
  Interventions: Other: Customized text message invitation ( Step 1a); Other: Customized automatic phone call invitation (Step 1b); Other: Secretary phone call (Step 2); Other: Health professional face-to-face appointment (Step 3)
- Written Letter (Active Comparator): Comparator will be the standard of care of invitation to cervical cancer screening: written letter
  Interventions: Other: Written Letter

INTERVENTIONS:
Other: Customized text message invitation ( Step 1a) — Personalized text messages, automatically sent by Smart Message v.3.1 software. These text messages intend to invite women to cervical cancer screening
  Arms: Stepwise intervention
Other: Customized automatic phone call invitation (Step 1b) — Personalized phone call, not operator dependent, automatically sent by Smart-Interactive Voice Response v.1.1 software These phone calls intend to invite women to cervical cancer screening
  Arms: Stepwise intervention
Other: Secretary phone call (Step 2) — Manual phone call, performed by a trained secretary. These phone calls invite women to cervical cancer screening, but will only be used after automatic strategies (customized text messages and phone calls)
  Arms: Stepwise intervention
Other: Health professional face-to-face appointment (Step 3) — Women randomized to experimental arm, who do not undergo cervical cancer screening after automatic invitation or manual phone call, receive this intervention. First, women are contacted through a phone call, performed by a health professional, inviting them for a face-to-face appointment at her primary care unit.
  During appointments, the health professional understands possible barriers felt by women for not undergoing cervical cancer screening. Health professionals will try to overcome these barriers, using pre-defined arguments and facts. Finally, women are invited to perform screening.
  Arms: Stepwise intervention
Other: Written Letter — A written letter will be used to invite eligible women to cervical cancer screening.
  This intervention will be used only for women randomized to active comparator arm.
  Arms: Written Letter

SUMMARY:
This study aims to assess the effectiveness of a stepwise approach, with increasing complexity and cost, to improve adherence to organized cervical cancer screening: step 1a - customized text message invitation; step 1b - customized automatic phone call invitation; step 2 - secretary phone call; step 3 - health professionals face-to-face appointment.

A population-based randomized controlled trial will be implemented in Portuguese urban and rural areas. Women eligible for cervical cancer screening will be randomized (1:1) to intervention and control. In the intervention group, women will be invited for screening through text messages, automatic phone calls, manual phone calls and health professional appointments, to be applied sequentially to participants remaining non-adherent after each step. Control will be the standard of care (invitation by written letter).

As primary objectives, we intend to test the superiority of interventions based on step 1 (1a+1b) and multistage interventions based on steps 1 and 2 and steps 1 to 3, based on intention-to-treat analyses.

DETAILED DESCRIPTION:
The secondary objectives will be the following:

1. To test the non-inferiority of interventions based on step 1a and step 1 (1a+1b), considering a non-inferiority limit of 5%;
2. To test the superiority of the specific components of the multistage intervention corresponding to step 2 and step 3;
3. To quantify the differences in adherence to cervical cancer screening, for interventions based on step 1 (1a+1b) and multistage interventions based on steps 1 and 2 and steps 1 to 3, between:

   1. Urban and rural areas;
   2. Younger and older population;
   3. Deprived and wealthy population;
   4. Never vs. ever users of screening;
   5. History of regular vs. irregular participation in screening programs.
4. To quantify the differences in adherence to cervical cancer screening when using a positive or a neutral content of text messages and automatic phone calls, in step 1;
5. To estimate the proportion of women who were performing cervical cancer screening in private health care services who started to be screened in an organized cervical cancer screening program, after a nurse face-to-face appointment at their primary care unit.

Intention-to-treat analysis will be used as primary strategy for all comparisons between interventions and control. Secondary per-protocol analysis will also be conducted. Binary logistic regression may be used to control for confounding, or in secondary analyses of the isolate effects of steps 1a, 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 25 and 49 years
* Medical registration at any of the primary health care units selected for this study
* Eligible for cervical cancer screening*

  * *Defined as all women aged between 25 and 60 years old who do not verify any of the following criteria: hysterectomized, active cervical cancer disease, currently undergoing cervical cancer treatment or did not start sexual activity.

Exclusion Criteria:

* Unavailability of mobile phone number

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1220 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Adherence to cervical cancer screening (step1) | Up to 20 months
  Proportion/cumulative proportion of women who performed cervical cancer screening on scheduled date, among those who were invited to undergo it, after step 1 or sequences of steps from 1 to 3

SECONDARY OUTCOMES:
Adherence to cervical cancer screening (steps 1a, 2 and 3) | Up to 20 months
  Proportion of women who performed cervical cancer screening on scheduled date, among those who were invited to undergo it, after step 1a, after step 2 or after step 3
Text message status | Up to 20 months
  Proportion of received text messages, from those that were sent
Automatic phone call status | Up to 20 months
  Proportion of delivered automatic phone calls, from those that were sent
Organized screening | Up to 20 months
  Proportion of women undergoing cervical cancer screening in a private health institution who changed to organized cervical cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Firmino DB Machado, MD, Principal Investigator — EPIUnit - Instituto de Saúde Pública da Universidade do Porto
Locations (2):
- Portugal (2):
  - ACeS Porto Ocidental, Porto
  - ACeS Marão e Douro Norte, Vila Real

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Firmino-Machado J, Varela S, Mendes R, Moreira A, Lunet N; SCAN-Cervical Cancer collaborators. A 3-step intervention to improve adherence to cervical cancer screening: The SCAN randomized controlled trial. Prev Med. 2019 Jun;123:250-261. doi: 10.1016/j.ypmed.2019.03.025. Epub 2019 Mar 30. PMID 30936001
- [Derived] Firmino-Machado J, Varela S, Mendes R, Moreira A, Lunet N; SCAN-Cervical Cancer collaborators. Stepwise strategy to improve cervical cancer screening adherence (SCAN-Cervical Cancer) - Automated text messages, phone calls and reminders: Population based randomized controlled trial. Prev Med. 2018 Sep;114:123-133. doi: 10.1016/j.ypmed.2018.06.004. Epub 2018 Jun 9. PMID 29894717
- [Derived] Firmino-Machado J, Mendes R, Moreira A, Lunet N. Stepwise strategy to improve Cervical Cancer Screening Adherence (SCAN-CC): automated text messages, phone calls and face-to-face interviews: protocol of a population-based randomised controlled trial. BMJ Open. 2017 Oct 5;7(10):e017730. doi: 10.1136/bmjopen-2017-017730. PMID 28982833